CLINICAL TRIAL: NCT05003999
Title: The Burden of Intermittent Catheterization in Adult Individuals With Neurogenic Lower Urinary Tract Dysfunction Following Spinal Cord Injury - Part 2
Brief Title: Time Needed to Perform Intermittent Catheterization in Adults With Spinal Cord Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrei Krassioukov (Other)
Collaborators: University of British Columbia (Other); International Collaboration on Repair Discoveries (Other); Vancouver Coastal Health (Other Government); Coloplast A/S (Industry)
Responsible Party: Sponsor-Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H17-03228 - Part 2; COLO-AK-NLUTD-SCI (Other Grant/Funding Number: Coloplast A/S)
Record Dates: First submitted 2021-06-22; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injuries; Neurogenic Lower Urinary Tract Dysfunction
Keywords: Spinal Cord Injury; Intermittent Catheterization; Hydrophilic Catheter; Non-Hydrophilic Catheter; Quality of Life; Time; Preparation; Satisfaction
MeSH Terms: conditions — Spinal Cord Injuries; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Two-by-two cross-over assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent catheterization starting with a hydrophilic catheter (HPC) (Experimental): The investigators measure the time taken to perform intermittent catheterization using a 13 step pre-determined intermittent catheterization protocol using a hydrophilic catheter i.e. SpeediCath ® (Coloplast A/S, Humlebæk, Denmark)
  Interventions: Device: HPC - SpeediCath ®
- Intermittent catheterization starting with a non-hydrophilic catheter (non-HPC) (Active Comparator): The investigators measure the time taken to perform intermittent catheterization using a 13 step pre-determined intermittent catheterization protocol using a non-hydrophilic catheter i.e. Self-Cath ® (Coloplast A/S, Humlebæk, Denmark); Lubrication jelly (MUKO ®, 3.5g package, Cardinal Health Canada Inc, Toronto, ON, Canada) was provided
  Interventions: Device: Non-HPC - Self-Cath ®

INTERVENTIONS:
Device: HPC - SpeediCath ® — The investigators measure the time taken to perform intermittent catheterization using a 13 step pre-determined intermittent catheterization protocol using a hydrophilic catheter
  Other Names: Intermittent catheterization using a hydrophilic catheter (HPC)
  Arms: Intermittent catheterization starting with a hydrophilic catheter (HPC)
Device: Non-HPC - Self-Cath ® — The investigators measure the time taken to perform intermittent catheterization using a 13 step pre-determined intermittent catheterization protocol using a non-hydrophilic catheter; Lubrication jelly (MUKO ®, 3.5g package, Cardinal Health Canada Inc, Toronto, ON, Canada) was provided
  Other Names: Intermittent catheterization using a non-hydrophilic catheter (non-HPC)
  Arms: Intermittent catheterization starting with a non-hydrophilic catheter (non-HPC)

SUMMARY:
This study investigates the burden of intermittent catheterization in adult individuals with neurogenic lower urinary tract dysfunction (NLUTD) following spinal cord injury (SCI).

Individuals will be recruited to compare two types of catheters. Each participant will use a non-hydrophilic catheter at one time point and a hydrophilic catheter at a different time point to perform intermittent catheterization. The order that participants use either a non-hydrophilic or a hydrophilic catheter will be determined randomly. The purpose of the study is to provide evidence for time spent on bladder management (performing intermittent catheterization) as well as consumer satisfaction on using both catheters.

DETAILED DESCRIPTION:
NLUTD and its management is of high priority for individuals living with SCI as it significantly reduces quality of life and interferes with their daily life. Intermittent catheterization in individuals with NLUTD following SCI is considered the preferred method of bladder emptying, i.e. gold standard.

Although intermittent catheterization offers reduced risk for urinary tract infection (UTI) compared to other methods of bladder emptying, the burden of complications including UTI and their management remains high. Another important aspect for individuals following SCI is improving quality of life. Since bladder management is a time-consuming and demanding task, reducing the time needed for intermittent catheterization and improving comfort during this procedure, i.e. convenience and ease of handling could significantly benefit quality of life for individuals living with SCI. Therefore, the investigators intend to compare hydrophilic versus non-hydrophilic catheters; time needed to perform intermittent catheterization and the convenience/ease of handling in this present study.

This is a prospective, randomized controlled crossover trial investigating the burden of intermittent catheterization in adult individuals with NLUTD following SCI.

Brief outline of study:

Visit 1 - Screening assessment to determine study eligibility. After providing informed consent, individuals will be assigned a unique study number and the following information will be collected:

* Inclusion / exclusion criteria
* Medical history including concomitant medication and procedures
* Demographic information

The following procedures will be conducted:

* Classification of SCI, i.e. neurological level and completeness using American Spinal Injury Association Impairment Scale (AIS)
* Participants will be randomized, i.e. either to start with the hydrophilic and non-hydrophilic catheter second or vice versa.

Visit 2 - Participants will perform intermittent catheterization to obtain a urine sample for culture (women will be administered a pregnancy test).

Visit 3 - Assessment of time to perform intermittent catheterization using catheter A or B (depending on randomization, e.g., starting with catheter A) followed by feedback on convenience and ease of handling using a satisfaction survey.

Visit 4 - Assessment of time to perform intermittent catheterization using catheter A or B (depending on randomization, e.g., now using catheter B) followed by feedback on convenience and ease of handling using a satisfaction survey.

Visit 5 - Individuals will receive a phone call and be asked to provide information regarding any changes in health and specifically bladder health.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* 18 years of age or older
* Presenting with a chronic SCI (i.e. greater than one year post-injury) at any level and with any severity (i.e. American Spinal Injury Association scale grade A to E )
* Hand function sufficient to perform intermittent catheterization for management of urinary bladder drainage
* Willing and able to comply with all clinic visits and study-related procedures
* Must provide informed consent and be able to understand and complete study-related instructions (must be able to understand and speak English)
* Women must not be pregnant
* Must not have any urinary diversion procedure, such as bladder augmentation, cystectomy, neo bladder, pouch reservoir, ileal conduit, Mitrofanoff appendicovesicostomy or similar

Exclusion Criteria:

* In addition to not fulfilling the inclusion criteria:

  * Presence of severe acute medical issue that in the investigator's judgement would adversely affect the individual's participation in the study
  * Individuals who do not perform intermittent catheterization
  * Individuals who are members of the investigational team and immediate family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Differences in time needed to perform intermittent catheterization between two types of catheters | Through study completion, an average of two weeks
  A measure of time (seconds) taken to perform intermittent catheterization using a 13 step pre-determined intermittent catheterization protocol where the first catheter will be different from the later catheter (i.e. hydrophilic vs. non-hydrophilic catheter).
Difference in convenience to perform intermittent catheterization between two types of catheters | Through study completion, an average of two weeks
  To assess the difference in convenience (ease of handling) for two catheters, i.e. using a hydrophilic vs. a non-hydrophilic catheter, as determined by using a survey.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD, PhD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ICORD is a spinal cord injury research centre of the UBC Faculty of Medicine and VCH Research Institute. — http://icord.org